CLINICAL TRIAL: NCT04898842
Title: BOUNCED: Managing Oral Diet Following a Diagnosis of Sub-acute Bowel Obstruction: a Feasibility Study Exploring the Efficacy of a 4 Stage Bowel Obstruction Cancer Diet and Quality of Life in Cancer Patients
Brief Title: Feasibility Study of a 4 Stage Bowel Obstruction Cancer Diet
Acronym: BOUNCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20DCSN272626
Record Dates: First submitted 2020-10-06; First posted 2021-05-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Adenocarcinoma; Colorectal Cancer Metastatic; Ovarian Cancer; Ovarian Neoplasm; Metastatic Colorectal Cancer; Metastatic Ovary Cancer; Peritoneal Carcinomatosis; Bowel Obstruction
Keywords: diet; dietary intervention
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Peritoneal Neoplasms; Intestinal Obstruction | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 stage bowel obstruction diet (Experimental): All eligible participants will be assessed by a specialist dietitian and a diet history and symptoms will be recorded. Depending on the degree of sub-acute bowel obstruction, symptoms and type of diet being followed, patients will be given detailed instructions on which stage of the 4 stage diet to use. They will be followed up by telephone or face to face weekly for a 4 week period and shown how to alter their diet by moving up and down the stage of the diet if symptoms resolve or worsen. This is current standard of care.
  Additional assessments will be carried out at the start and end of the study when participants will complete the Memorial Symptom Assessment Scale (MSAS) and EORTC QLQ-30 quality of life questionnaire. They will be asked to complete a daily diet diary, and an 'ease of use' questionnaire at the end of the 4 week period.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — To determine whether a 4 stage bowel obstruction diet as a means of managing oral intake in patients symptomatic with malignant sub-acute bowel obstruction (SBO) is deliverable and effective in clinical practice.

SUMMARY:
Bowel obstruction is a common complication in patients with ovarian, peritoneal and bowel cancer due to a mass or spread of disease, causing narrowing to the gut, as these cancers can grow on the bowel surface. Certain foods may lead to symptoms such as pain, bloating, feeling full, feeling sick, vomiting and difficulty passing a bowel motion.

There is limited evidence to establish the best diet to follow when someone is diagnosed with the risk of bowel obstruction and is experiencing symptoms after eating and drinking.

The Dietitians at the Royal Surrey have developed a 4 stage bowel obstruction diet which they have been using with patients for 3 years. The 4 stages are clear fluids, all thin liquids, low fibre soft smooth diet, low fibre soft sloppy diet. Depending on the severity of symptoms and the risk of a blockage, patients are asked to follow a certain stage of the diet. They are advised to move up and down the stages as symptoms improve or get worse.

This feasibility study aims to investigate if the diet can be used and is effective in clinical practice. The objectives are to see if this diet is easy to follow, can reduce symptoms of bowel obstruction, can improve quality of life, and reduce admissions to hospital because of bowel blockages.

Patients at risk of bowel obstruction from colorectal or ovarian cancer are eligible to participate. They will remain in the study for a period of 4 weeks, during which time they will be asked to complete a diet diary and 3 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Able to tolerate oral diet
* Confirmed diagnosis of SBO due to underlying malignancy to include:

  1. Patients with colorectal or gynaecological cancers with primary or secondary tumour in situ, undergoing cancer treatment or supportive care.
  2. Patients diagnosed with advanced inoperable cancers of colorectal or gynaecological origin
* Presenting in outpatient clinics or admitted from A&E with a minimum of 2 symptoms of SBO including: abdominal pain, bloating after eating, early satiety, nausea, vomiting
* Capacity to give informed consent

Exclusion Criteria:

* Patients under 18 years of age
* No symptoms of bowel obstruction
* Have not already been given advice to follow the 4 stage bowel obstruction diet
* Unable to tolerate oral diet i.e. enterally or parenterally fed
* Unable to provide capacity to give informed consent
* Unable to read and communicate in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Symptoms of sub-acute bowel obstruction: abdominal pain, feeling bloated, feeling full-up quickly, nausea and / or vomiting | 4 weeks
  Measured by completion of the Memorial Symptom Assessment Scale questionnaire (MSAS): a well-validated questionnaire, which asks about the frequency, severity and psychological effect of 32 symptoms. For the purpose of this study, the MSAS has been adapted to include the key additional symptom of early satiety (feeling full up quickly) that can be experienced by patients with sub-acute bowel obstruction. It is graded on a scale of 0 (not at all) - 4 (very much).

SECONDARY OUTCOMES:
A&E attendances or hospital admissions after starting to use the 4 stage diet | 4 weeks
  No of hospital admissions and A&E attendances due to bowel obstruction in the 3 months prior to consent will be recorded. This will be compared with the number of admissions during the 4 weeks patients are on the trial.
Health related Quality of Life | 4 weeks
  Measured by using the EORTC Quality of Life QLQ-C30 questionnaire will be collected at baseline on entry to the study and after 4 weeks on completion of the study. QLQ-C30 developed by EORTC is designed to measure cancer patients' physical, psychological and social functions. It is scored on a scale from 0 (not at all) - 4 (very much).
Weight | 4 weeks
  Measured in kilograms and as a percentage indicating percentage weight change from start to end of the trial. Participants will be weighed on consent and after 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Allan, Principal Investigator — Royal Surrey NHS Foundation Trust; Agnieszka Michael, Principal Investigator — Royal Surrey NHS Foundation Trust
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No